CLINICAL TRIAL: NCT05114590
Title: A 16-week, Multicenter, Prospective, Open-label, Single-arm, Phase 4 Study to Evaluate the Effect of Soliqua™ 100/33 on the Percentage of Time in Range (TIR) From Continuous Glucose Monitoring (CGM) in Insulin-naïve Patients With Very Uncontrolled Type 2 Diabetes Mellitus
Brief Title: Effect of Soliqua 100/33 on Time in Range From Continuous Glucose Monitoring in Insulin-naive Patients With Very Uncontrolled Type 2 Diabetes Mellitus
Acronym: Soli-CGM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16990; U1111-1261-7399 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- iGlarLixi (Experimental): iGlarLixi (i.e., insulin glargine 100 Units/ml /lixisenatide 33 μg/mL) once daily for 16 weeks.
  Interventions: Drug: Insulin glargine/Lixisenatide

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide — Solution for injection in a pre-filled pen by subcutaneous injection. Dose was individually titrated to achieve target fasting self-monitoring of plasma glucose (SMPG) of 80 to 100 milligrams per deciliter (mg/dL) (4.4 to 5.6 millimoles per liter [mmol/L]) while avoiding hypoglycemia.
  Other Names: iGlarLixi; Soliqua 100/33; AVE0010-1

SUMMARY:
The purpose of the study was to demonstrate if iGlarLixi (Soliqua 100/33) would improve glycemic control (as measured by Time in Range) and glycemic variability in participants with very uncontrolled (HbA1c ≥ 9%) type 2 Diabetes Mellitus (T2DM) while on at least 2 oral antidiabetic drugs [OADs] with or without a glucagon-like peptide 1 receptor agonist [GLP1 RA]), as measured by continuous glucose monitoring (CGM).

The total study duration per participant was approximately 22 weeks. Three site visits, 3 site or home visits, and up to 13 phone contacts were scheduled.

* A screening period of up to 2 weeks
* A run-in period of up to 2 weeks, including the baseline period
* A 16-week, open-label treatment period
* A 2-week post-treatment safety follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes mellitus (T2DM) for at least 6 months before the baseline period
* HbA1c ≥9-13% during the run-in period
* On at least 2 OADs with or without GLP-1 RA with stable doses (for both) for 3 months prior to the screening period
* Willing and able to wear the CGM device continuously for 14 days to capture CGM measures at baseline until the next site visit and again towards the end of the treatment period
* Willing and able to prick fingers a minimum of 2-4 times per week utilizing sterile lancets provided along with a manual blood glucose meter kit
* Willing to discontinue the daily (oral or injectable) or weekly GLP-1 RA or DPP 4i prior to administration of iGlarLixi (Soliqua 100/33)
* Willing and able to inject iGlarLixi (Soliqua 100/33) and increase dose as needed to achieve SMPG target
* Non-pregnant, non-breastfeeding women utilizing a highly-effective contraceptive method or of non-childbearing potential

Exclusion Criteria:

* Type1 Diabetes mellitus (T1DM) or any other types of diabetes, except T2DM
* On meglitinides (eg, nateglinide, repaglinide)
* Body mass index (BMI) >40 kg/m² during the screening period
* Any current or previous skin conditions, including (but not limited to) severe psoriasis, burns, eczema, scarring, excessive tattoos, that would inhibit the proper wearing of the CGM device
* History of severe nausea and vomiting leading to subsequent discontinuation of GLP-1 RA
* Known history or presence of clinically significant pancreatitis or gastroparesis
* Participants with an episode of severe hypoglycemia or with hypoglycemia unawareness (defined as the onset of neuroglycopenia before the appearance of autonomic warning symptoms [for example, blurred vision, difficulty speaking, feeling faint, difficulty thinking, and confusion] or as the failure to sense a significant fall in blood glucose below normal levels) diagnosed within the 6 months prior to the screening period
* Participants with personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predisposed to MTC (eg, multiple endocrine neoplasia syndromes)
* Significant current (within past 2 months) and/or expected use of medications known to affect glycemia (eg, ≥5 mg/day prednisone)
* Use of substances known to interfere with CGM readings, such as aspirin-containing products (>650 mg/day of salicylic acid) or supplements containing vitamin C (>1000 mg/day of ascorbic acid) during the 14 days of CGM at either baseline or end of treatment period
* Previous treatment with any insulin (except for short term treatment due to intercurrent illness, including gestational diabetes, at the discretion of the investigator)
* Had used weight loss drugs (including over the counter and herbal medications) within 12 weeks before the screening visit

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- United States (18):
  - Clearview Medical Research LLC-Site Number:8400003, Canyon Country, California
  - National Research Institute - ClinEdge - PPDS-Site Number:8400004, Huntington Park, California
  - National Research Institute - ClinEdge - PPDS-Site Number:8400009, Huntington Park, California
  - Torrance Clinical Research Institute-Site Number:8400008, Lomita, California
  - Downtown LA Research Center Inc - ClinEdge - PPDS-Site Number:8400001, Los Angeles, California
  - University Clinical Investigators Inc-Site Number:8400020, Tustin, California
  - San Fernando Valley Health Institute - ClinEdge - PPDS-Site Number:8400012, West Hills, California
  - Premier Research Associate-Miami-Site Number:8400002, Miami, Florida
  - Floridian Research Institute-Site Number:8400013, Miami, Florida
  - Palm Research Center, Inc.-Site Number:8400005, Las Vegas, Nevada
  - Hassman Research Institute - HRI - Berlin - CenExel - PPDS-Site Number:8400007, Berlin, New Jersey
  - Mid Hudson Medical Research PLLC-Site Number:8400014, New Windsor, New York
  - Endocrinology Associates Inc-Site Number:8400011, Columbus, Ohio
  - University of Tennessee Health Science Center-Site Number:8400017, Memphis, Tennessee
  - University of Texas Southwestern Medical Center-Site Number:8400018, Dallas, Texas
  - Flourish Research - San Antonio - PPDS-Site Number:8400006, San Antonio, Texas
  - Northeast Clinical Research of San Antonio LLC-Site Number:8400019, Schertz, Texas
  - Consano Clinical Research LLC-Site Number:8400010, Shavano Park, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16990 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25293&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centers in the United States. A total of 244 participants were screened between 27 January 2022 and 03 December 2022, of which 120 were screen failures. Screen failures were mainly due to not meeting glycated hemoglobin inclusion criteria.
Pre-assignment Details: A total of 124 participants were enrolled in the study.
Groups:
- iGlarLixi: Participants received iGlarLixi (Soliqua 100/33) subcutaneous injection once daily for 16 weeks.
Period: Overall Study
Arm/Group | iGlarLixi
Started | 124
Completed the 16-week Study Treatment Period | 111
Completed (Completed study per protocol.) | 110
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Investigator decision | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 5
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Enrolled set included all eligible participants who were dispensed iGlarLixi and signed the informed consent form.
Groups:
- iGlarLixi: Participants received iGlarLixi subcutaneous injection once daily for 16 weeks.
Arm/Group | iGlarLixi
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6
  Black | 21
  White | 89
  Multiple | 1
  Not Reported | 2
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in the Percentage of Time in Range [70 to 180 Milligram Per Deciliter (mg/dL)]
Description: The percentage of time spent in the glycemic target range of 70 to 180 mg/dL was calculated as 100 times the number of recorded measurements in the glycemic target range (70 to 180 mg/dL inclusive), divided by the total number of recorded measurements. Baseline is defined as the first 14 evaluable days of evaluable continuous glucose monitoring (CGM) data prior to first day of treatment. CGM compliance is defined as 1) at least 8 out of 14 days (not necessarily consecutive) have 100% of evaluable CGM data per 24-hour period (at least 8 days with 96 records minimum per day) OR 2) at least 9 out of 14 days (not necessarily consecutive) have ≥89% of evaluable CGM data per 24-hour period (at least 9 days with 85 records minimum per day) OR 3) at least 10 out of 14 days (not necessarily consecutive) have at least ≥80% of evaluable CGM data per 24 hour period (at least 10 days with 77 records minimum per day).
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: Efficacy analysis set included all enrolled participants who received >=1 dose of iGlarLixi and had evaluable CGM data at baseline. Only participants analyzed at baseline and Week 16 are reported.
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | iGlarLixi
Number analyzed (Participants) | 113
percentage of time | 26.22 [20.5 to 31.9]

2. Secondary Outcome: Percent Change From Baseline to Week 16 in Glucose Total Coefficient of Variation (CV)
Description: Glucose total CV was calculated by following: standard deviation glucose/mean glucose over 14 days x 100, and the percent change was reported. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of treatment.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | iGlarLixi
Number analyzed (Participants) | 113
percent change | 5.0 [3.8 to 6.1]

3. Secondary Outcome: Change From Baseline to Week 16 in Mean Daily Blood Glucose
Description: A global average was computed to determine the average of the mean daily blood glucose for the 14 days at baseline and Week 16. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of treatment.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | iGlarLixi
Number analyzed (Participants) | 113
mg/dL | -52.48 [-64.6 to -40.3]

4. Secondary Outcome: Change From Baseline to Week 16 in the Maximum Postprandial Glucose Exposure in the 4 Hours Post-Breakfast Meal
Description: The analysis was focused on the 4-hour interval at both baseline and Week 16 from t=0 (the timepoint at which glucose measurement was taken immediately preceding liquid meal administration) throughout the subsequent 4 hours. For each participant, the overall maximum glucose value within the described 4-hour period was determined, and the difference between the maximum glucose value at baseline and Week 16 was reported. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of treatment.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | iGlarLixi
Number analyzed (Participants) | 118
mg/dL | -73.66 [-90.9 to -56.4]

5. Secondary Outcome: Change From Baseline to Week 16 in Time Above Range (>180 mg/dL)
Description: The time spent above the glycemic target range was calculated as 100 times the total number of 15-minute increments of CGM data where a participant's blood glucose falls above normal range (>180 mg/dL) at baseline, divided by the total number of 15-minute increments read (i.e., up to 1344 15-minute increments) at Week 16. This was calculated for baseline and Week 16 and the change was reported. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of treatment.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | iGlarLixi
Number analyzed (Participants) | 113
percentage of time | -28.67 [-34.6 to -22.7]

6. Secondary Outcome: Percentage of Participants Who Achieved Coefficient of Variation <36%
Description: Percentage of participants achieving CV <36% was calculated as sum of the number of participants with CV <36% divided by the total number of participants. The endpoint was calculated using all CGM glucose readings available throughout each day for 2 weeks (Week 14-16).
Time Frame: Week 16
Population: Efficacy analysis set included all enrolled participants who received >=1 dose of iGlarLixi and had evaluable CGM data at baseline. Only participants analyzed at Week 16 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iGlarLixi
Number analyzed (Participants) | 100
percentage of participants | 76.0 [66.4 to 84.0]

7. Secondary Outcome: Change From Baseline to Week 16 in Time in Range Per Time Blocks
Description: Time spent in the glycemic target range (70 to 180 mg/dL) was calculated as 100 times the number of recorded measurements in the glycemic target range (70 to 180 mg/dL inclusive), divided by the total number of recorded measurements per time block and comparing the corresponding time blocks from Week 16 to baseline. The time blocks are 12 am to 6 am, 6 am to 12 pm, 12 pm to 6 pm, 6 pm to 12 am, and 6 am to 12 am. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of treatment.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of time
Arm/Group | iGlarLixi
Number analyzed (Participants) | 100
percentage of time
  12 am to 6 am | 27.89 [21.3 to 34.5]
  6 am to 12 pm | 33.73 [27.0 to 40.5]
  12 pm to 6 pm | 31.05 [24.5 to 37.6]
  6 pm to 12 am | 25.87 [19.8 to 31.9]
  6 am to 12 am | 30.21 [24.1 to 36.3]

8. Secondary Outcome: Percentage of Participants Who Achieved Glucose Management Indicator (GMI) <7% and <9%
Description: The GMI was calculated as 3.31 + 0.02392 x (mean glucose in mg/dL from CGM data). The GMI was calculated by determining the number of participants who achieved <7% and <9% at Week 16.
Time Frame: Week 16
Population: Efficacy analysis set included all enrolled participants who received >=1 dose of iGlarLixi and had evaluable CGM data at baseline. Only participants with GMI data available at Week 16 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iGlarLixi
Number analyzed (Participants) | 100
percentage of participants
  GMI <7% | 43.0 [33.1 to 53.3]
  GMI <9% | 85.0 [76.5 to 91.4]

9. Secondary Outcome: Change From Baseline to Week 16 in the 4-Hour Postprandial Glucose Area Under the Concentration Time Curve From 0 to 4 Hours
Description: Blood samples were collected to measure the glucose values up to 4-hour after the breakfast meal. The analysis was based on a liquid meal at both baseline and Week 16 (a liquid meal administered in a fasted state and blood glucose is measured at specific time points up to 4 hours). Baseline is defined as the time period prior to administration of study drug.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL*hour
Arm/Group | iGlarLixi
Number analyzed (Participants) | 102
mg/dL*hour | -325.93 [-390.6 to -261.2]

10. Secondary Outcome: Change From Baseline to Week 16 in Time to Reach Maximum Postprandial Glucose Concentration
Description: Blood samples were collected at specific intervals over a 4 hour period to measure blood glucose values following ingestion of a liquid meal and the process is repeated after 16 weeks of study drug administration following another liquid meal administration and blood glucose values measured at specific time points over 4 hours. The difference in the time to reach the maximal blood glucose value was then calculated between these two timepoints.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: hour
Arm/Group | iGlarLixi
Number analyzed (Participants) | 103
hour | -0.24 [-0.5 to 0.0]

11. Secondary Outcome: Percentage of Participants Who Spent <15 Minutes/Day at a Glucose Level <54 mg/dL
Description: Blood glucose level was determined based upon CGM data. Percentage of participants with glucose level <54 mg/dL for less than 15 minutes per day are reported.
Time Frame: Week 16
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iGlarLixi
Number analyzed (Participants) | 100
percentage of participants | 63.0 [52.8 to 72.4]

12. Secondary Outcome: Change From Baseline to Week 16 in Overall Score of Diabetes Medication Treatment Satisfaction Scores Using the Diabetes Medication Satisfaction Tool (DM-SAT) Questionnaire
Description: The changes in diabetes medication treatment-related impact and satisfaction was measured by the DM-SAT. The DM-SAT is a 16-item measure with 4 domains/subscales assessing lifestyle (5 items), medical control (3 items), convenience (5 items) and well being (3 items). Each item is measured on a scale from 0-10, where 0= not at all satisfied, 1 to 3= not too satisfied, 4 to 6 = somewhat satisfied, 7-9= very satisfied and 10= extremely satisfied. The overall score was calculated as the sum of the 16 questions with a score that ranges from 0 to 160. A higher score indicates a positive result. Baseline is defined as the first 14 evaluable days of evaluable CGM data prior to first day of administration.
Time Frame: Baseline (Days -14 to -1) and Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | iGlarLixi
Number analyzed (Participants) | 106
units on a scale | 0.18 [0.14 to 0.22]

13. Secondary Outcome: Number of Participants With Confirmed Hypoglycemia Measured by Blood Glucose Levels
Description: Hypoglycemia event is defined as any event recorded in hypoglycemic event information library electronic case report form page that has "Yes" as the response to the question "Were any hypoglycemic events experienced".
  American Diabetes Association (ADA) Level 1 hypoglycemia is defined as measurable glucose concentration <70 mg/dL [3.9 millimoles per liter (mmol/L)] but >=54 mg/dL (3.0 mmol/L).
  ADA Level 2 hypoglycemia is defined as measurable glucose concentration <54 mg/dL (3.0 mmol/L) that needed immediate action.
  ADA Level 3 hypoglycemia is defined as severe event characterized by altered mental and/or physical functioning that required assistance from another person for recovery of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest.
  Participants might have experienced both Level 1 and 2 hypoglycemia events.
Time Frame: From the first administration of the study drug (Day 1) up to 3 days after last administration of the study drug (maximum exposure duration: up to 16 weeks)
Population: Safety set included all enrolled participants who received >=1 dose of iGlarLixi.
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi
Number analyzed (Participants) | 123
Participants
  Any Hypoglycemia events | 35
  Hypoglycemia events confirmed by ADA criteria | 29
  ADA Level 1 hypoglycemia | 26
  ADA Level 2 hypoglycemia | 11
  ADA Level 3 hypoglycemia | 0

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, whether or not considered related to the study drug. An SAE is defined as any AE that, at any dose, meets one of the following criteria: results in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity or congenital anomaly/birth defect. TEAEs is defined as AEs that developed, worsened, or became serious during the treatment-emergent period, defined as the time from the first administration of the study drug (Day 1) to the last administration of the study drug + 3 days.
Time Frame: as for outcome 13
Population: Safety set included all enrolled participants who received >=1 dose of iGlarLixi.
Measure: Count of Participants; unit: Participants
Arm/Group | iGlarLixi
Number analyzed (Participants) | 123
Participants
  Any TEAE | 47
  Any treatment-emergent SAE | 1

ADVERSE EVENTS:
Time Frame: TEAEs data was collected from the first administration of the study drug (Day 1) up to 3 days after last administration of the study drug (maximum exposure duration: up to 16 weeks).
Description: Analysis was performed on the safety set.
Arm/Group | iGlarLixi
All-Cause Mortality (participants affected / at risk) | 0/123
Serious Adverse Events (participants affected / at risk) | 1/123
Other Adverse Events (participants affected / at risk) | 14/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iGlarLixi (N=123)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iGlarLixi (N=123)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05114590/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05114590/SAP_001.pdf